CLINICAL TRIAL: NCT03568604
Title: Open-Label Vulvoscopy Photography Study of Changes in Vulva, Vestibule, Urethral Meatus and Vagina 20 Weeks Post Daily Administration of 6.5 Mg Vaginal Prasterone in Menopausal Women With Moderate to Severe Dyspareunia
Brief Title: Changes to Vulva, Vestibule, Urethral Meatus and Vagina 20 Weeks Post Daily Prasterone in Women With Dyspareunia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Diego Sexual Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDSM-2018-01
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Dyspareunia
Keywords: vulvovaginal atrophy; dyspareunia; prasterone; vulvoscopy
MeSH Terms: conditions — Dyspareunia | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: Open label study of daily administration of 6.5 mg prasterone, approved for moderate to severe dyspareunia for vaginal atrophy in menopausal women, to see if there are changes to the vulva, vestibule, urethral meatus and vagina on vulvoscopy after 20 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prasterone (Experimental): 6.5 mg vaginal inserts of prasterone will be used daily once the patient meets inclusion and exclusion for 20 weeks.
  Interventions: Drug: Prasterone

INTERVENTIONS:
Drug: Prasterone — 6.5 vaginal insert prasterone (dehydroepiandrosterone)
  Other Names: Intrarosa

SUMMARY:
Open label study at a single research center. Subjects meeting inclusion and exclusion criteria will receive 6.5 mg prasterone vaginal inserts daily for twenty weeks. A physical examination and vulvoscopy with photography of the vulva, vestibule, urethral meatus and vagina will be performed at baseline and every 4 weeks for 20 weeks. Pain diaries will be completed between visits.

DETAILED DESCRIPTION:
This is an open label study to be conducted at a single research center, San Diego Sexual Medicine. Subjects meeting inclusion and exclusion criteria will receive 6.5 mg prasterone vaginal inserts daily for twenty weeks. After the informed consent is signed, a baseline physical examination and vulvoscopy with detailed photography of the vulva, vestibule, urethral meatus and vagina will be performed. Physical examination and vulvoscopy with detailed photography of the vulva, vestibule, urethral meatus and vagina will be repeated prospectively every 4 weeks for a total of 20 weeks. Therefore, physical examination and vulvoscopy with detailed photography of the vulva, vestibule, urethral meatus and vagina will be performed prospectively at baseline (vulvoscopy session 1), 4 weeks (vulvoscopy session 2), 8 weeks (vulvoscopy session 3), 12 weeks (vulvoscopy session 4), 16 weeks (vulvoscopy session 5) and 20 weeks (vulvoscopy session 6) following daily administration of 6.5 mg prasterone. In addition, pain diaries will be dispensed at each visit and collected at the following visit, with questions regarding pain during sexual activity.

ELIGIBILITY:
Inclusion Criteria:

* provides written informed consent and HIPAA authorization before any study procedures are conducted;
* has a body mass index (BMI) < 37 kg/m2
* is menopausal either naturally (at least 12 months amenorrheic) or 6 weeks after a bilateral salpingo-oophorectomy prior to natural menopause; subjects with hysterectomy only must have a serum FSH > 40 mIU/mL;
* has vulvovaginal atrophy with moderate to severe dyspareunia;
* has at least one score ≥ 2 on cotton-tipped swab test
* agrees to comply with the study procedures and visits.

Exclusion Criteria:

* has a hypersensitivity to DHEA;
* has used prasterone in the past 6 months;
* has documented or suspected breast cancer;
* has undiagnosed genital bleeding:
* has clinically significant findings on physical examination;
* has uncontrolled hypertension;
* has any chronic medical condition or psychologic disorder that the Principal Investigator feels makes her ineligible for the study;
* is currently on local or systemic androgen therapy including local or systemic testosterone (washout 14 days for local or topical androgen or non-depot injection, 1 month for depot, 6 months for pellet;
* is currently on local or systemic estrogen therapy or androgen therapy (washout 14 days for vaginal estrogen, 60 days for oral/transdermal therapy);
* is currently using a selective estrogen receptor modulator (SERM) or products that have estrogenic or anti-estrogenic effects within last month;
* has a history of substance abuse within 12 months prior, or consuming > 14 alcoholic drinks per week;
* has received an investigational drug within 30 days prior to signing consent;
* has any condition or exhibits behavior that indicates to the Principal Investigator that the Subject is unlikely to be compliant with study procedures and visits.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Vulvoscopic changes to the vulva, vestibule, urethral meatus and vaginal region on VGTA scale | Twenty weeks
  The primary objective of this study is to prospectively document, using vulvoscopy with detailed photography, the visible changes to the vulva, vestibule, urethral meatus and vaginal region in menopausal women with moderate to severe dyspareunia using 6.5 mg daily prasterone for twenty weeks, comparing baseline to 20 weeks. Photographs will be assessed by an independent reviewer using a ten-parameter Likert rating scale, the Vulvoscopic Genitourinary Tissue Appearance (VGTA) scale. This scale assesses for labia majora resorption, labia minora resorption, clitoral atrophy, urethral meatal prolapse, introital stenosis, pallor, erythema, mucosa inflammation, loss of vaginal ruggation, and anterior vaginal wall atrophy. VGTA values for each parameter are 0 (normal), 1(mild), 2 (moderate) or 3 (severe). Each parameter will be calculated separately as well as the total score as primary outcome measure.

SECONDARY OUTCOMES:
Changes in pain as noted on cotton-tipped swab (Q-tips®) test. | Twenty weeks
  Secondary objectives include changes in pain as noted on the Pain Scale during the cotton-tipped swab (Q-tips®) test. Pain is assessed by applying pressure with the cotton-tipped swab in 7 specific locations around the vestibule (1:00, 3:00, 5:00, 6:00, 7:00, 9:00 and 11:00) and the patient is asked to assess her pain at each location on a scale of 0-3 with 0 being no pain and 3 being the most severe. The total score is then used to determine outcome.
Subject diary | Twenty weeks
  Changes in responses to questions on subject diary from first 4 week period prior to start of medication, to last 4 week period ending at twenty weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, MD, Principal Investigator — San Diego Sexual Medicine; Sue W Goldstein, BA, CCRC, Study Director — San Diego Sexual Medicine
Locations (1):
- San Diego Sexual Medicine, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Background] Labrie F, Archer DF, Martel C, Vaillancourt M, Montesino M. Combined data of intravaginal prasterone against vulvovaginal atrophy of menopause. Menopause. 2017 Nov;24(11):1246-1256. doi: 10.1097/GME.0000000000000910. PMID 28640161
- [Background] Labrie F, Martel C. A low dose (6.5 mg) of intravaginal DHEA permits a strictly local action while maintaining all serum estrogens or androgens as well as their metabolites within normal values. Horm Mol Biol Clin Investig. 2017 Feb 1;29(2):39-60. doi: 10.1515/hmbci-2016-0042. PMID 27997350
- [Background] Martel C, Labrie F, Archer DF, Ke Y, Gonthier R, Simard JN, Lavoie L, Vaillancourt M, Montesino M, Balser J, Moyneur E; other participating members of the Prasterone Clinical Research Group. Serum steroid concentrations remain within normal postmenopausal values in women receiving daily 6.5mg intravaginal prasterone for 12 weeks. J Steroid Biochem Mol Biol. 2016 May;159:142-53. doi: 10.1016/j.jsbmb.2016.03.016. Epub 2016 Mar 10. PMID 26972555
- [Background] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686
- [Background] Bouchard C, Labrie F, Derogatis L, Girard G, Ayotte N, Gallagher J, Cusan L, Archer DF, Portman D, Lavoie L, Beauregard A, Cote I, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Group. Effect of intravaginal dehydroepiandrosterone (DHEA) on the female sexual function in postmenopausal women: ERC-230 open-label study. Horm Mol Biol Clin Investig. 2016 Mar;25(3):181-90. doi: 10.1515/hmbci-2015-0044. PMID 26725467
- [Background] Labrie F, Derogatis L, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; Members of the VVA Prasterone Research Group. Effect of Intravaginal Prasterone on Sexual Dysfunction in Postmenopausal Women with Vulvovaginal Atrophy. J Sex Med. 2015 Dec;12(12):2401-12. doi: 10.1111/jsm.13045. Epub 2015 Nov 23. PMID 26597311
- [Background] Archer DF, Labrie F, Bouchard C, Portman DJ, Koltun W, Cusan L, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Treatment of pain at sexual activity (dyspareunia) with intravaginal dehydroepiandrosterone (prasterone). Menopause. 2015 Sep;22(9):950-63. doi: 10.1097/GME.0000000000000428. PMID 25734980
- [Background] Labrie F, Archer D, Bouchard C, Fortier M, Cusan L, Gomez JL, Girard G, Baron M, Ayotte N, Moreau M, Dube R, Cote I, Labrie C, Lavoie L, Gilbert L, Martel C, Balser J. Lack of influence of dyspareunia on the beneficial effect of intravaginal prasterone (dehydroepiandrosterone, DHEA) on sexual dysfunction in postmenopausal women. J Sex Med. 2014 Jul;11(7):1766-85. doi: 10.1111/jsm.12517. Epub 2014 Apr 28. PMID 24774442
- [Background] Labrie F, Martel C, Berube R, Cote I, Labrie C, Cusan L, Gomez JL. Intravaginal prasterone (DHEA) provides local action without clinically significant changes in serum concentrations of estrogens or androgens. J Steroid Biochem Mol Biol. 2013 Nov;138:359-67. doi: 10.1016/j.jsbmb.2013.08.002. Epub 2013 Aug 14. PMID 23954500